CLINICAL TRIAL: NCT01517711
Title: A Double-Blind, Placebo-Controlled, Flexible-Dose Pilot Clinical Trial of Once-Daily Extended-Release Tramadol for the Treatment of PTSD
Brief Title: Tramadol Extended-Release (ER) for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INTRuST-Tramadol
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: pharmacotherapy; combat disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tramadol ER (Experimental): Tramadol in an extended release formulation with an initial dosage of 100 mg daily, increased weekly over the next two weeks, as tolerated, to a maximum of 300 mg daily
  Interventions: Drug: Tramadol
- Placebo capsule (Placebo Comparator): Lactose encapsulated to match appearance of experimental drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol — Tramadol hydrochloride Extended Release(ER) will be supplied as tablets of Ultram® ER 100mg. Tramadol ER (100-300mg) or matching placebo will be self-administered by oral route every morning (with or without food) for 6 weeks. Patients will be instructed to take it the same way (either with food or without food) each time they take their dose. Each patient will be provided with 1 week supply of Tramadol ER or matching placebo on visits 2 (week 0) and 3 (week 1) and 2 weeks supply on visits 4 (week 2) and 5 (week 4).
  Other Names: Ultram® ER
  Arms: Tramadol ER
Drug: Placebo — Matching placebo will be self-administered by oral route every morning (with or without food) for 6 weeks. Patients will be instructed to take it the same way (either with food or without food) each time they take their dose. Each patient will be provided with 1 week supply of Tramadol ER or matching placebo on visits 2 (week 0) and 3 (week 1) and 2 weeks supply on visits 4 (week 2) and 5 (week 4).
  Arms: Placebo capsule

SUMMARY:
This was a six-week pilot study testing the efficacy of tramadol extended-release (ER) for posttraumatic stress disorder (PTSD). Men and women aged 21-55 years with combat-related PTSD or PTSD resulting from a civilian trauma were recruited. Blinded tramadol ER was begun with a 100 mg daily dose for the first week, with an option to increase to 200 mg/day for the 2nd week. Dose adjustments, using a range of 100-300 mg tramadol ER per day (or 1 to 3 placebo tabs), were permitted thereafter. The primary hypothesis was that tramadol ER 100 to 300 mg every morning for 6 weeks would reduce the symptoms of PTSD relative to placebo. The primary outcome measures were PTSD symptoms as rated by the Clinician-Administered PTSD Scale (CAPS) and Clinicians Global Impressions scale at baseline and weeks one, two, four, and six.

DETAILED DESCRIPTION:
This was a single-site, double-blind, placebo-controlled, randomized, 6-week, parallel-group, flexible-dose outpatient trial of tramadol ER 100-300 mg once every morning for PTSD. Double-blinded clinical outcome measures were obtained during screening, and at weeks 0 (pre-randomization), 1, 2, 4, and 6; outcome was also assessed at week 7, the follow-up and study discharge visit, which occurred one week after the discontinuation of study medicine. Tramadol ER (or placebo) was started at 100 mg daily and increased weekly over the next two weeks, as tolerated, to a maximum of 300 mg daily. Dose change was also permitted at week 4. Matching drug and placebo were prepared by a research pharmacy using over-encapsulation in locking DB capsules supplied by Capsugel. Lactose was used as a filler to attain uniformity in weight. Randomization used a 1:1 allocation ratio and was via a block design, with stratification by military service. Other than the research pharmacists, all study personnel, all staff, and all subjects were blind.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, military veterans and non-veterans, aged 21-55 years
2. Active PTSD as determined by diagnostic evaluation and standardized interview (Structured Clinical Interview for the DSM (SCID))
3. Literacy and ability to give informed consent
4. In women of child-conceiving potential, a negative pregnancy test and use of an approved birth control method
5. Glasgow Coma Scale (GCS) score of 15, Extension of GCS with 7-point Amnesia Scale score of 6 (amnesia for traumatic event of 30 min or fewer) or 7 (no amnesia for impact of head) (Nell et al 2000)
6. Clinically judged to be at low risk for adverse sequelae from taking tramadol
7. Concomitant medications must be approved by the PI

Exclusion Criteria:

1. Pregnant or nursing women
2. Homeless persons
3. Suicidal or homicidal ideation with plans or intent
4. History of opioid dependence or abuse
5. Psychosis or history thereof, substance dependence or abuse (other than tobacco dependence; lifetime opioid abuse is exclusionary) within the past 60 days, anorexia nervosa, antisocial personality disorder, or other psychiatric disorder judged by the investigator to be more clinically significant than PTSD
6. Serious or unstable illness, endocrinopathy, or metabolic instability, including renal insufficiency, liver disease, hydrocephalus, history of stroke, history of seizures, history of brain tumor
7. Use of non-study medications except those approved by the PI
8. Newly started in psychotherapy (< 3months)
9. History of hypersensitivity, allergy, or other significant adverse effects from tramadol

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Geracioti, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Cincinnati VA Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Geracioti TD. Tramadol treatment of combat-related posttraumatic stress disorder. Ann Clin Psychiatry. 2014 Aug;26(3):217-21. PMID 25166484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 subjects were consented to achieve sample of 40; one never returned for evaluation.
Pre-assignment Details: 40 evaluable subjects
Period: Overall Study
Arm/Group | Tramadol ER | Placebo
Started | 22 | 18
Completed | 20 | 15
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol ER | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.7) | 33.7 (7.0) | 32.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 20 | 13 | 33
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The Clinician-Administered PTSD Scale (CAPS) is an interview-based measure of severity of PTSD symptoms. A total score is calculated with a range of 0-136, with higher numbers indicating more severe symptoms.
Time Frame: Weeks 0 (baseline),1, 2, 4, 6
Population: 33 men and 7 women with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tramadol ER Men; Tramadol ER Women: Tramadol: Tramadol hydrochloride Extended Release(ER) will be supplied as tablets of Ultram® ER 100mg. Tramadol ER (100-300mg) or matching placebo will be self-administered by oral route every morning (with or without food) for 6 weeks. Patients will be instructed to take it the same way (either with food or without food) each time they take their dose. Each patient will be provided with 1 week supply of Tramadol ER or matching placebo on visits 2 (week 0) and 3 (week 1) and 2 weeks supply on visits 4 (week 2) and 5 (week 4).
- Placebo Men; Placebo Women: Placebo: Matching placebo will be self-administered by oral route every morning (with or without food) for 6 weeks. Patients will be instructed to take it the same way (either with food or without food) each time they take their dose. Each patient will be provided with 1 week supply of Tramadol ER or matching placebo on visits 2 (week 0) and 3 (week 1) and 2 weeks supply on visits 4 (week 2) and 5 (week 4).
Arm/Group | Tramadol ER Men | Placebo Men | Tramadol ER Women | Placebo Women
Number analyzed (Participants) | 20 | 13 | 2 | 5
units on a scale
  Week 0 | 79.1 (17.8) | 81.9 (24.8) | 90.0 (5.7) | 91.0 (19.0)
  Week 1 | 62.5 (24.7) | 69.8 (25.0) | 68.5 (10.6) | 71.0 (24.3)
  Week 2 | 54.4 (25.7) | 68.5 (26.2) | 67.0 (31.1) | 62.2 (15.4)
  Week 4 | 46.4 (30.2) | 61.0 (28.4) | 39.5 (55.9) | 47.0 (14.3)
  Week 6 | 46.5 (32.2) | 51.0 (28.6) | 36.0 (50.9) | 41.0 (14.4)
Statistical Analysis 1: Comparison: Tramadol ER Men vs Placebo Men; Women were excluded from analysis because of the small sample size and unequal distribution across groups; Test type: Superiority or Other; p = 0.286, ANOVA — P value is for overall post-randomization CAPS score

2. Primary Outcome: Clinical Global Impression -- Improvement (CGI-I) -- Subject
Description: The Clinicial Global Impression - Improvement (CGI-I) is a single item rated by a clinician. The range is 1 (very much improved)) to 7 (very much worse).
Time Frame: Week 6, assessing clinician's judgment of change from week 0 to week 6
Population: 33 men and 7 women with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol ER Men | Placebo Men | Tramadol ER Women | Placebo Women
Number analyzed (Participants) | 20 | 13 | 2 | 5
units on a scale | 2.3 (1.1) | 2.6 (1.1) | 2.0 (1.4) | 1.6 (0.5)
Statistical Analysis 1: Comparison: Tramadol ER Men vs Placebo Men; Test type: Superiority or Other; p < 0.10, ANOVA

3. Secondary Outcome: Visual Analog Scales (VAS)
Description: Self-rated 100-mm visual analog scales [0 to 100 scale; higher score indicates more of the rated state] to rate poor sleep, happiness, irritability, nervousness and pain. Change is calculated by subtracting week 6 from week 0.
Time Frame: Change from week 0 to 6
Population: 33 men and 7 women with PTSD
Measure: Mean (Standard Deviation); unit: change in mm
Groups:
- Tramadol Men; Tramadol Women: Tramadol: Tramadol hydrochloride Extended Release(ER) will be supplied as tablets of Ultram® ER 100mg. Tramadol ER (100-300mg) or matching placebo will be self-administered by oral route every morning (with or without food) for 6 weeks. Patients will be instructed to take it the same way (either with food or without food) each time they take their dose. Each patient will be provided with 1 week supply of Tramadol ER or matching placebo on visits 2 (week 0) and 3 (week 1) and 2 weeks supply on visits 4 (week 2) and 5 (week 4).
Arm/Group | Tramadol Men | Placebo Men | Tramadol Women | Placebo Women
Number analyzed (Participants) | 20 | 13 | 2 | 5
change in mm
  Poor sleep | 26.8 (38.5) | 6.7 (31.5) | 51.0 (31.1) | 32.8 (14.1)
  Happiness | -18.5 (33.4) | -11.0 (27.3) | -40.3 (2.5) | -29.6 (42.2)
  Irritability | 18.0 (30.5) | 14.2 (39.4) | 52.5 (16.3) | 39.0 (22.4)
  Nervousness | 15.0 (31.9) | 9.5 (24.3) | 34.0 (5.7) | 36.4 (26.9)
  Pain | 7.5 (22.8) | 10.4 (21.3) | 41.0 (1.4) | 5.6 (31.8)
Statistical Analysis 1: Comparison: Tramadol Men vs Placebo Men; Analysis is for sleep only (men); Test type: Superiority or Other; p = 0.03, ANOVA

4. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS)
Description: Quick Inventory of Depressive Symptoms - Self Report (QIDS) is a self-report scale of severity of depression. A total score is calculated with a range of 0 to 27, with higher numbers indicating greater severity.
Time Frame: Weeks 0, 1, 2, 4 and 6
Population: 33 men and 7 women with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol Men | Placebo Men | Tramadol Women | Placebo Women
Number analyzed (Participants) | 20 | 13 | 2 | 5
units on a scale
  QIDS week 0 | 11.2 (4.2) | 13.7 (4.4) | 15.5 (2.1) | 12.6 (4.8)
  QIDS week 1 | 8.7 (4.8) | 11.8 (4.2) | 11.0 (5.7) | 8.4 (4.2)
  QIDS week 2 | 7.7 (4.7) | 11.6 (5.6) | 12.0 (9.9) | 7.0 (2.2)
  QIDS week 4 | 7.7 (5.6) | 10.0 (5.2) | 9.0 (8.5) | 7.1 (4.6)
  QIDS week 6 | 6.7 (4.8) | 7.1 (4.1) | 6.5 (4.9) | 4.5 (1.7)

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Adverse events were assessed via study measures and clinician interview.
Arm/Group | Tramadol ER | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 7/22 | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol ER (N=22) | Placebo (N=18)
Headache (Nervous system disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes